CLINICAL TRIAL: NCT02039037
Title: Efficacy of Acupuncture and Electroacupuncture in Patients With Chronic Nonspecific Low Back Pain: Randomized Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, JOSIELLI COMACHIO, Efficacy of Acupuncture and Electroacupuncture in patients with chronic nonspecific low back pain: randomized clinical trial, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: josicomachio
Record Dates: First submitted 2013-10-30; First posted 2014-01-17 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Acupuncture Therapy; Electroacupuncture

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acupuncture group (Active Comparator): This group perform acupuncture needles brand Dong Bang 20x15 in specific spots for the treatment of low back pain.
  Interventions: Device: Acupuncture
- Electroacupuncture group (Active Comparator): Electro Group, will be added through the use of electrical stimulation of electroacupuncture using the apparatus Accurate pulse 585 at the same points.
  Interventions: Device: Electroacupuncture (device 585)

INTERVENTIONS:
Device: Acupuncture — Acupuncture Group, which will hold acupuncture needles brand Dong Bang 20x15 in specific spots for the treatment of low back pain.
  Arms: Acupuncture group
Device: Electroacupuncture (device 585) — Electro will be added through the use of electrical stimulation to the Electro Accurate use of the device 585 at the same points Pulse.
  Arms: Electroacupuncture group

SUMMARY:
Chronic nonspecific low back pain is a major health and socioeconomic responsible for a high rate of employee absenteeism and reduced functional performance. The use of acupuncture as an alternative therapy in the treatment of low back pain and electroacupuncture to enhance the treatment has been effective; however, there is little evidence of the effectiveness of one over the other.

DETAILED DESCRIPTION:
OBJECTIVE: To compare the effect of acupuncture and electroacupuncture as an alternative therapy in patients with chronic low back pain to be able to identify whether electroacupuncture has more benefits than just acupuncture in the treatment of low back pain to be more widespread with scientific.

METHOD: Sixty subjects will be randomized into two groups: Group Acupuncture treatment of low back pain (AG) and Group Acupuncture with the use of electroacupuncture (EG). The primary clinical outcomes will be pain, assessed with the numerical pain scale and McGill Pain Questionnaire and disability assessed with Roland Morris Disability Questionnaire. Secondary outcomes will be measured with global perception scale of global perceived effect, quality of life using the Short-Form Health Survey questionnaire (SF-36), Beck Depression (Beck Depression Inventory BDI), Flexibility, kinesiophobia and through bank Wells. The groups will be treated with two weekly sessions lasting about an hour, 6 weeks, totaling 12 sessions. The outcomes will be achieved in the final and initial ratings after six months of treatment completion. Data will be collected by a blinded examiner who also has made the allocation of patients to groups.

ELIGIBILITY:
Inclusion Criteria:

* Chronic low back pain (pain for more than three months)
* Be between 20-60 years

Exclusion Criteria:

* Patients with severe spinal
* Previous surgeries or scheduled
* Herniated Disc
* Rheumatic disease or infection
* pregnancy
* metal implants

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Pain | 6 weeks
  Pain Numerical Rating Scale (NRS) and McGill Pain Questionnaire
Functional Disability | 6 weeks
  Roland Morris Disability Questionnaire

SECONDARY OUTCOMES:
Scale of Kinesiophobia (TSK) | 6 weeks
  Self-applied questionnaire of 17 items, which was developed to measure the fear of movement due to cLBP. Each question has 4 4 response options (strongly disagree, agree, and strongly agree) with scores respectively ranging from 1 to 4 points.
Quality of life | 6 weeks
  Short-Form Health Survey Questionnaire
Global Perceived Effect | 6 weeks
  Global Perceived Effect Scale
Beck Depression | 6 weeks
  Beck Depression Inventory BDI
Third finger to the ground | 6 weeks
  Third finger of the hand to the ground test to assess the flexibility of the posterior chain.

CONTACTS AND LOCATIONS:
Overall Officials: Josielli Comachio, Principal Investigator — University of Sao Paulo
Locations (1):
- Medicine School of the University Of São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Comachio J, Oliveira Magalhaes M, Nogueira Burke T, Vidal Ramos LA, Peixoto Leao Almeida G, Silva AP, Ferreira de Meneses SR, Costa-Frutuoso JR, Santos Miotto Amorim C, Pasqual Marques A. Efficacy of acupuncture and electroacupuncture in patients with nonspecific low back pain: study protocol for a randomized controlled trial. Trials. 2015 Oct 15;16:469. doi: 10.1186/s13063-015-0850-7. PMID 26472590